CLINICAL TRIAL: NCT06926946
Title: The Effects of Treatment Guided by Cerebral Oximetry Monitoring on Renal Outcomes in Invasively Mechanically Ventilated Neonates: an Ancillary Study of the SafeBoosC-IIIv Trial
Brief Title: SafeBoosC-IIIv - Does Cerebral Oximetry Monitoring Affect Renal Outcomes
Acronym: SBIIIvR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: St. John's Research Institute (Other)
Collaborators: Rigshospitalet, Denmark (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 229/2024
Record Dates: First submitted 2025-04-02; First posted 2025-04-15 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Acute Renal Failure; Neonatal Morbidity
Keywords: Cerebral oximetry; NIRS; Neonate; Ventilated; Kidney injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Arm- Cerebral Oximetry + Treatment Guideline (Experimental): Neonates who are ventilated in the NICU, in addition to standard care, will be monitored by cerebral oximetry. If the value falls below a certain threshold, the treatment guideline will be followed and corrective interventions undertaken.
  Interventions: Other: Intervention Arm- Cerebral Oximetry + Treatment Guideline
- Control Arm- standard care (No Intervention): Neonates who are ventilated in the NICU will receive standard care only.

INTERVENTIONS:
Other: Intervention Arm- Cerebral Oximetry + Treatment Guideline — if the cerebral oximeter shows low values, a pre designed treatment guideline will be followed and corrective actions taken.
  Other Names: NIRS
  Arms: Intervention Arm- Cerebral Oximetry + Treatment Guideline

SUMMARY:
Cerebral oximetry monitoring allows clinicians to optimize blood flow to the brain and oxygenation using the SafeBoosC treatment guideline. The guideline's interventions aims to stabilize blood pressure and oxygen levels.

As low blood pressure is a risk factor for the development of kidney injury, normalizing blood pressure may decrease the incidence of kidney injury in new-borns who are on ventilator.

ELIGIBILITY:
Inclusion Criteria:

* > 28 weeks of gestation Invasively ventilated

Exclusion Criteria:

* major anomalies

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1000 (Estimated)
Dates: Start 2025-07-31 (Estimated); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-09-15 (Estimated)

PRIMARY OUTCOMES:
composite outcome of death and acute kidney injury | From randomization to discharge up to 2months of life
  composite outcome of death and acute kidney injury

CONTACTS AND LOCATIONS:
Locations (1):
- St. jOhn's Medical college & Hospital, Bengaluru, Karnataka, India

IPD SHARING:
Plan to Share IPD: No